CLINICAL TRIAL: NCT03554512
Title: TelePremie: Telehomecare for Step-down Care Post-NICU Discharge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Horizon Health Network (Other)
Collaborators: Canada Health Infoway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHSTHCHHN02
Record Dates: First submitted 2018-05-04; First posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-05

CONDITIONS: Anxiety; Self Efficacy
Keywords: Neonatal Intensive Care; Telehealth; Anxiety; Self Efficacy; Parenting/psychology
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): No Intervention
- Telehealth (Experimental): Telehealth virtual appointment
  Interventions: Other: Telehealth virtual appointment

INTERVENTIONS:
Other: Telehealth virtual appointment — Appointment with NICU clinician via telehealth equipment.
  Arms: Telehealth

SUMMARY:
Telehealth is a means of providing care from a distance, at the convenience of the patient. This study will be testing the addition of Telehealth visits (TH) to the standard of care (SOC) following discharge from the neonatal intensive care unit (NICU). This study will be used to determine whether Telehealth appointments post-NICU discharge can improve the experiences of parents in caring for their infant and reduce the number of health care visits they have with their infant within three months post-NICU discharge.

Participants in this study will be randomly assigned to two groups. One group will receive the standard of care, which means they will have an appointment in place with a primary care provider, pediatrician or return visit to the NICU post discharge. The second group will have the standard of care described above and two Telehealth visits within the first week at home with their infant.

The study will explore the experiences of parents of NICU infants following their discharge from NICU, both those receiving standard of care (SOC) and the Telehealth monitoring intervention. Participants will be required to complete surveys online at 5 time periods: when parents decide to be part of the study, prior to discharge from NICU, 1 day after discharge, 2 days following the primary care provider visit and at 3 months following discharge from NICU. The questionnaires used will measure parental anxiety levels and parental confidence. The number of infant visits to the primary care provider, pediatrician, emergency department and NICU will also be collected at three months post-NICU discharge.

A subset of participants (from both SOC and TH groups) will further participate in semi-structured interviews about their experiences in the NICU and caring for their children after discharge. NICU clinicians who consent will participate in semi-structured interviews about their experiences with the Telehealth intervention.

The cost-effectiveness of the Telehealth intervention will be analysed in comparison to SOC.

ELIGIBILITY:
Inclusion Criteria:

* Parent-infant pairs admitted to neonatal intensive care unit where study is conducted.
* Parent has internet access.
* Parent has literacy level such that they are comfortable reading and filling out surveys.
* Infant is likely to survive.

Exclusion Criteria:

* Infant discharged to foster care.
* Infant transferred or discharged within 3 days of admission to neonatal intensive care unit.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
The State-Trait Anxiety Inventory | Change from Baseline State-Trait Anxiety at 3 months
The Maternal Confidence Questionnaire | Change from Baseline self-efficacy at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Cecil Ojah, MD, Principal Investigator — Horizon Health Network
Locations (1):
- Saint John Regional Hospital, Saint John, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No